CLINICAL TRIAL: NCT01444482
Title: A Phase I Single Blinded Randomised Exploratory Trial in Elderly Volunteers to Assess and Compare Safety and Immunogenicity of Adjuvanted Seasonal Influenza Vaccine (Investigational Vaccine) to Standard Seasonal Influenza Vaccine.
Brief Title: Study of Parenterally Administrated Adjuvanted Seasonal Influenza Vaccine in Healthy Elderly Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Isconova AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ISC-Influenza-001
Record Dates: First submitted 2011-08-19; First posted 2011-09-30 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Matrix-M

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Matrix M adjuvanted influenza vaccine (Experimental): 1 human dose of seasonal influenza vaccine formulated with 50 µg Matrix M
  Interventions: Biological: Matrix M
- Seasonal influenza vaccine (Active Comparator): 1 human dose of seasonal influenza vaccine
  Interventions: Biological: Seasonal influenza vaccine

INTERVENTIONS:
Biological: Matrix M — 1 human dose of seasonal influenza vaccine formulated with 50 µg Matrix M, total dosage volume 0.55 mL injected intramuscularly in the upper arm once at day 0.
  Arms: Matrix M adjuvanted influenza vaccine
Biological: Seasonal influenza vaccine — 1 human dose of seasonal influenza vaccine
  Arms: Seasonal influenza vaccine

SUMMARY:
The safety of parenterally administrated investigational vaccine (commercial influenza vaccine formulated with adjuvant Matrix M) in healthy adults (age 18-50) and healthy elderly (age 65-75), will be investigated in the study. Moreover, the study aims to study parameters associated with improved protection against clinical disease in elderly. Such parameters include HI-titres, a balanced Th1/Th2 response as well as a functional cellular immune response.

Vaccination will start in 22 healthy adults receiving the investigational vaccine. Vaccination of elderly will be initiated only after demonstration of safety in adults. 88 healthy elderly volunteers will be vaccinated, 44 will receive the seasonal influenza vaccine alone and 44 will receive the investigational vaccine. Vaccines will be administrated intramuscularly in the upper arm. One dose will be administered to each volunteer included in the study. Blood samples for basic immunological assessments of cellular and humoral immunity will be taken at day 0, 7, 28, 90 and 150.

The investigational vaccine is equal to one standard human dose of a commercial seasonal influenza vaccine to which 50 µg of adjuvant Matrix M has been added.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 18 to 50 years for the young adult part of the study
* Are aged 65 to 75 years for main study
* Have signed a voluntary written informed consent. Volunteers should be cooperative, willing and able to participate and adhere to the Protocol requirements
* Have minimum normal standard physical performance status

Exclusion Criteria:

* Volunteer has received seasonal Influenza vaccine of same antigenic composition within 6 months prior to enrolment
* Volunteer having vaccine specific HI titres ≥ 40
* Volunteer is taking immunosuppressant drugs such as azathioprine, tacrolimus, cyclosporine, etc
* Volunteers who have primary or secondary immunodeficiencies (e.g. Human Immunodeficiency Virus [HIV])
* Volunteers who have an autoimmune disease
* Volunteer is taking oral, intramuscular or intravenous corticosteroids. Use is not permitted within 1 month of Screening. Inhaled corticosteroids to treat respiratory insufficiency (e.g. chronic obstructive pulmonary disease [COPD]), are permitted
* Volunteer has a concurrent severe or uncontrolled underlying medical disease unrelated but that is likely to compromise volunteer safety and affect the outcome of the study
* Volunteer has a neurotoxicity (Grade ≥2)
* Volunteer has diarrhoea (Grade ≥2)
* Volunteer has received other vaccines, within 1 month prior to enrolment
* Volunteer has a history of any severe or life-threatening hypersensitivity reaction
* Volunteer has an unstable systemic disease (including active infection, uncontrolled hypertension [> 160/100], unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal and metabolic disease)
* Volunteer has recent history (within 6 months) of chronic alcohol or drug abuse of which may compromise the patient's safety or ability to participate in study activities
* Volunteer has a history of psychiatric disorder that prevents patients from providing informed consent or following Protocol instructions
* Volunteer is currently enrolled in an investigational device or drug trial, or < 1 month since completing an investigational device or drug trial
* Female volunteers who are pregnant or lactating (only applicable for Pre-Study)
* Volunteer has any other factor that in the opinion of the Investigator (or designee) would make the patient unsafe or unsuitable for the study

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Safety in elderly and adults given a single parenterally administrated dose of seasonal influenza vaccine adjuvanted with Matrix M | 1 - 3 months

SECONDARY OUTCOMES:
Immunogenicity in adults and elderly given a dose of seasonal influenza vaccine adjuvanted with Matrix M | 1 - 7 months
Immunogenicity in elderly given a dose of seasonal influenza vaccine alone or adjuvanted with Matrix M | 1 - 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Drug Reseach Center, Balatonfüred, Balatonfured, Hungary